CLINICAL TRIAL: NCT06574724
Title: Transfer of Microorganisms Between Green Areas and Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Irina Spacova, Prof., Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B3002024000110
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-08

CONDITIONS: Microbial Colonization
Keywords: green areas; nature; microbiome; biodiversity; sequencing
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Green space intervention (Experimental): Participants that visit a green space
  Interventions: Other: Visiting a green space

INTERVENTIONS:
Other: Visiting a green space — Participants are asked to visit a green space for a defined time period

SUMMARY:
The goal of this study is to understand how visiting green areas affects the human microbiome through microbial transfer. Additionally, the project aims to understand which environmental, health and lifestyle factors can influence these microbiome changes. Participants will visit a green area, provide microbiome samples before and after the visit, and complete questionnaires related to environmental, health, lifestyle and demographic factors.

DETAILED DESCRIPTION:
Several hypotheses propose that the modern surge in immune disorders is related to diminished contact with nature. Specifically, the Biodiversity hypothesis emphasizes that contact with natural environments enriches the human microbiome and is necessary for promoting immune balance. This project aims to investigate whether visiting green areas can contribute to changes in human microbiome composition. Additionally, the investigators aim to explore the environmental, health and lifestyle factors that can influence these microbiome changes. Adults and/or children will be asked to visit a green space (such as an urban park) and perform specific activities (such as walking or pushing a stroller) for a defined time period. Before and after this visit, swabs of their skin and nose will be collected to analyze microbiome changes. In addition, questionnaires will be administered to the participants, with the goal to align microbiome changes with environmental, health, lifestyle and demographic factors.

ELIGIBILITY:
Inclusion criteria:

Children (min. 4 years old) and adult participants (18+) of any gender in generally good health.

No strict exclusion criteria will be set in advance.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2027-07-07 (Estimated); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
Microbiome changes | Two time points directly before and after the intervention (on 1 day)
  Microbiome sequencing will be performed to assess changes in microbial community composition of nasal and skin swabs, focusing on abundances and diversity of different microorganisms and their genes

SECONDARY OUTCOMES:
Specific microorganisms within the skin and nasal microbiomes | Two time points directly before and after the intervention (on 1 day)
  Specific microorganisms within the participants' microbiomes will be assessed through culturing of swabs and/or quantification via qPCR
Associations between the human microbiome and environment | Two time points directly before and after the intervention (on 1 day)
  Human microbiome composition and diversity (as assessed in outcome "Microbiome changes") will be correlated with the green space environment characteristics, such as the environmental (microbiome) biodiversity

OTHER OUTCOMES:
Self-reported lifestyle | One time point directly before or after the intervention (on 1 day)
  Lifestyle will be assessed using a short questionnaire to understand how it might impact the microbiome (as assessed in outcome "Microbiome changes"), reflecting lifestyle-related parameters such as weekly time spent outdoors (in hours) and frequency of exposure to green environments (e.g., once a year)
Self-reported health | One time point directly before or after the intervention (on 1 day)
  Self-reported general health will be assessed using a short questionnaire to understand how it might impact the microbiome (as assessed in outcome "Microbiome changes"), reflecting health-related parameters such as a health rating (from very poor to very good)
Self-reported demographic information | One time point directly before or after the intervention (on 1 day)
  Demographic information will be assessed using a short questionnaire to understand how it might impact the microbiome (as assessed in outcome "Microbiome changes"), reflecting demographic parameters such as age (in years), gender, and parent-child relationship (having one or more children)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Spacova, Prof., Principal Investigator — Universiteit Antwerpen; Stijn Verhulst, Prof. dr., Principal Investigator — Universiteit Antwerpen and University Hospital Antwerp (UZA)
Locations (1):
- Universiteit Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No